CLINICAL TRIAL: NCT05188677
Title: A Multi-center, Observer-blind, Randomized, Controlled Phase 3 Study to Evaluate the Immunogenicity and Safety of Adjuvanted Recombinant SARS-CoV-2 Trimeric S-protein Subunit Vaccine (SCB-2019), Administered as a Booster Dose to Adults, Who Previously Received Primary Series of a COVID-19 Vaccine
Brief Title: Immunogenicity and Safety Study of SCB-2019 Vaccine as a Booster to COVID-19 Vaccine in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Clover Biopharmaceuticals AUS Pty (Industry)
Responsible Party: Sponsor
Organization: Clover Biopharmaceuticals, Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CLO-SCB-2019-015
Record Dates: First submitted 2022-01-10; First posted 2022-01-12 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — SCB-2019 COVID-19 vaccine; ChAdOx1 nCoV-19; sinovac COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Group 1a (primary series: Comirnaty) (Experimental): participants will receive one dose of SCB-2019 vaccine on Day 1
  Interventions: Biological: Candidate vaccine, SCB-2019
- Group 1b (primary series: Comirnaty) (Active Comparator): participants will receive one dose of Comirnaty vaccine on Day 1
  Interventions: Biological: Comirnaty Vaccine
- Group 2a (primary series: Vaxzevria) (Experimental): participants will receive one dose of SCB-2019 vaccine on Day 1
  Interventions: Biological: Candidate vaccine, SCB-2019
- Group 2b (primary series: Vaxzevria) (Active Comparator): participants will receive one dose of Vaxzevria vaccine on Day 1
  Interventions: Biological: Vaxzevria Vaccine
- Group 3a (primary series: CoronaVac) (Experimental): participants will receive one dose of SCB-2019 vaccine on Day 1
  Interventions: Biological: Candidate vaccine, SCB-2019
- Group 3b (primary series: CoronaVac) (Active Comparator): participants will receive one dose of CoronaVac vaccine on Day 1
  Interventions: Biological: CoronaVac Vaccine
- Group 4a (primary series and booster dose CoronaVac) (Experimental): participants will receive one dose of SCB-2019 vaccine on Day 1
  Interventions: Biological: Candidate vaccine, SCB-2019
- Group 4b (primary series and booster dose CoronaVac) (Active Comparator): participants will receive one dose of CoronaVac on Day 1;
  Interventions: Biological: CoronaVac Vaccine
- Group 4c (primary series and booster dose CoronaVac) (Experimental): participants will receive a half dose of SCB-2019 vaccine on Day 1
  Interventions: Biological: Candidate vaccine, SCB-2019
- Group 5a (primary series: CoronaVac) (Experimental): participants will receive a dose of 2-vial presentation of SCB-2019 vaccine
  Interventions: Biological: Candidate vaccine, SCB-2019
- Group 5b (primary series: CoronaVac) (Experimental): participants will receive a dose of 3-vial presentation of SCB-2019 vaccine
  Interventions: Biological: Candidate vaccine, SCB-2019

INTERVENTIONS:
Biological: Candidate vaccine, SCB-2019 — a recombinant SARS-CoV-2 trimeric S-protein subunit vaccine for COVID-19; intramuscular injection
  Arms: Group 1a (primary series: Comirnaty); Group 2a (primary series: Vaxzevria); Group 3a (primary series: CoronaVac); Group 4a (primary series and booster dose CoronaVac); Group 4c (primary series and booster dose CoronaVac); Group 5a (primary series: CoronaVac); Group 5b (primary series: CoronaVac)
Biological: Comirnaty Vaccine — intramuscular injection
  Arms: Group 1b (primary series: Comirnaty)
Biological: Vaxzevria Vaccine — intramuscular injection
  Arms: Group 2b (primary series: Vaxzevria)
Biological: CoronaVac Vaccine — intramuscular injection
  Arms: Group 3b (primary series: CoronaVac); Group 4b (primary series and booster dose CoronaVac)

SUMMARY:
The purpose of this study is to assess the immunogenicity and safety of the investigational SCB-2019 vaccine, administered as a booster dose, to adults who:

* Received primary series with one of the selected authorized or investigational COVID-19 vaccines at least 3 months prior to enrollment.
* Received primary series and a booster dose of CoronaVac at least 3 months prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants at least 18 years of age;
* Individuals willing and able to comply with study requirements, including all scheduled visits, vaccinations, laboratory tests, and other study procedures;
* Individuals willing and able to give an informed consent, prior to screening;
* Healthy participants or participants with pre-existing medical conditions who are in a stable medical condition;
* Individuals who received primary vaccination series with one of the selected COVID-19 vaccines (Comirnaty, Vaxzevria, or CoronaVac) ≥3 months prior to enrollment; or received primary series and a booster dose (≥3 months after primary series) of CoronaVac, ≥3 months prior to enrollment.

Exclusion Criteria:

* Individuals with fever >37.5°C (axillary), or any acute illness at baseline (Day 1) or within 3 days prior to randomization;
* Individuals with laboratory-confirmed SARS-CoV-2 infection at Visit 1 (determined by positive Rapid Antigen Test or RT-PCR);
* Individuals who have received an investigational or licensed COVID-19 vaccine prior to Day 1 (except for primary series with Comirnaty, Vaxzevria, CoronaVac vaccines, or primary and booster dose of CoronaVac), or plan to receive COVID-19 vaccine during the study period;
* Individuals who have a history of severe adverse reaction associated with a vaccine or severe allergic reaction (e.g., anaphylaxis) to any component of the study vaccines;
* Individuals who have received any other investigational product within 30 days prior to Day 1 or intend to participate in another clinical study at any time during the conduct of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1831 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
GMT ratio of GMT SCB-2019 over GMT Comirnaty on Day 15 | Day 15
GMT ratio of GMT SCB-2019 over GMT COVID-19 Vaccine Janssen on Day 15 | Day 15
GMT ratio of GMT SCB-2019 over GMT CoronaVac Vaccine on Day 15 | Day 15
Local and systemic solicited AEs reported within 7 days after study vaccination | Up to 7 days after each vaccination
Unsolicited AEs reported from Visit 1 (Day 1) through Safety Call Day 29 | Up to Day 29
SAEs, AEs leading to early termination from the study, MAAEs, and AESIs | Through study completion, an average of 6 Months

CONTACTS AND LOCATIONS:
Locations (2):
- Philippines (2):
  - Las Piñas Doctors Hospital, Las Piñas, National Capital Region
  - Manila Doctors Hospital, Manila, National Capital Region

REFERENCES:
- [Derived] Roa CC Jr, de Los Reyes MRA, Plennevaux E, Smolenov I, Hu B, Gao F, Ilagan H, Ambrosino D, Siber G, Clemens R. Superior Boosting of Neutralizing Titers Against Omicron SARS-CoV-2 Variants by Heterologous SCB-2019 Vaccine vs a Homologous Booster in CoronaVac-Primed Adults. J Infect Dis. 2023 Nov 2;228(9):1253-1262. doi: 10.1093/infdis/jiad262. PMID 37439701